CLINICAL TRIAL: NCT06026124
Title: Retrieval-Based Word Learning in Developmental Language Disorder During Book Reading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Laurence Leonard, Professor of Speech, Language, & Hearing Sciences, Purdue University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1603017480C; R01DC014708 (NIH)
Record Dates: First submitted 2023-08-11; First posted 2023-09-06 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Developmental Language Disorder; Specific Language Impairment; Language Development
Keywords: word learning; word retrieval; preschool-aged children
MeSH Terms: conditions — Language Development Disorders; Specific Language Disorder

STUDY DESIGN:
Intervention Model Description: Within-participant design in which each child learns words under two conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Developmental Language Disorder (Experimental): These children have a significant delay in language development in the absence of hearing impairment, cognitive delay, autism, or neurological injury/disease.
  Interventions: Behavioral: Retrieval-based word learning: Repeated Spaced Retrieval condition; Behavioral: Retrieval-based word learning: Repeated Study condition
- Children with typical language development (Experimental): Children whose language development is as expected for their age.
  Interventions: Behavioral: Retrieval-based word learning: Repeated Spaced Retrieval condition; Behavioral: Retrieval-based word learning: Repeated Study condition

INTERVENTIONS:
Behavioral: Retrieval-based word learning: Repeated Spaced Retrieval condition — Each child will learn 8 novel nouns referring to unfamiliar plants and animals ("nepp") and a related "meaning" ("a nepp likes rain") in the context of a story book. Four of the nouns will be will be learned using repeated spaced retrieval. In this condition, they will initially hear the information and be asked to retrieve it. Thereafter, they will be asked to retrieve it after hearing 3 intervening words. After each retrieval attempt, they will hear the target information again. This procedure will occur on two consecutive days.
Behavioral: Retrieval-based word learning: Repeated Study condition — Each child will learn 8 novel nouns referring to unfamiliar plants and animals ("nepp") and a related "meaning" ("a nepp likes rain") in the context of a story book. Four of the nouns will be will be learned using repeated study trials only (with no retrieval practice). In this condition, they will simply hear the information (word & meaning) as part of the story. This procedure will occur on two consecutive days.

SUMMARY:
Children with developmental language disorder (DLD; also referred to as specific language impairment) experience a significant deficit in language ability that is longstanding and harmful to the children's academic, social, and eventual economic well-being. Word learning is one of the principal weaknesses in these children. This project focuses on the word learning abilities of four- and five-year-old children with DLD. The goal of the project is to build on the investigators' previous work to determine whether, as has been found thus far, special benefits accrue when these children must frequently recall newly introduced words during the course of learning. In this study, the investigators seek to replicate the advantage that repeated retrieval holds over simple exposure to the words and to demonstrate an increase in children's absolute levels of learning by implementing retrieval practice in the context of a story book.

DETAILED DESCRIPTION:
Developmental Language Disorder (DLD) affects language learning in an estimated 7% of children. Although much of the research literature has emphasized difficulties learning grammar, children with DLD also have major deficits in vocabulary. In recent work, the investigators have been examining the benefit of retrieval practice to enhance word learning and retention in preschoolers with DLD. The rationale behind this work is grounded in the growing literature in the field of cognitive psychology which shows that repeated practice in retrieving information results in greater long-term retention than continuous study of that information without opportunities for retrieval. In addition, retrieval practice that occurs after a delay-or "spacing" between study of a word and subsequent recall attempts-can lead to stronger effects.

The investigators have explored the benefits of retrieval practice for preschoolers with DLD and with typical language development (TD), showing that recall and retention for novel words (nouns, adjectives, verbs) were greater when learned using repeated spaced retrieval (RSR) than when learned using repeated study only. Despite benefitting from RSR, children with DLD still showed lower levels of recall than children with TD.

In the current study, the investigators aim to increase accuracy levels by embedding the same words and retrieval schedules used in earlier studies into story contexts. Artist-illustrated stories incorporate illustrations of the unfamiliar plants and animals that served as referents of novel nouns in an earlier study. Sixteen children with DLD will be recruited for this study along with 16 children with TD matched on chronological age. Using a within-subjects design, children will learn eight novel nouns, four embedded in each story. Along with each word form, children will learn a "meaning", that is, an additional piece of semantic information about the referent.

For words in the RSR condition, each novel word and meaning, paired with its referent, will be presented as part of the story. Immediately after hearing it, children will be asked to recall both form and meaning, and then will hear those repeated. All subsequent retrieval trials will occur after three other words have intervened since the last time the word appeared in a study trial. Novel words assigned to the comparison condition will simply be heard paired with their referent during the story at the same frequency as words in the RSR condition. Children will not be asked to recall the words in the comparison condition during the learning period. Stories will be presented twice on each of the learning days. As written, the stories are a reasonable length and pace, but by repeating the story, children will hear the words the same number of times overall as in the investigator's previous studies, allowing evaluation of the benefits of the story format. Recall of the word forms and meanings will be tested after the story book reading on the second day and one week later. One week later, the recall test will be re-administered and children will complete a three-alternative recognition test.

The investigators hypothesize that children will show greater recall for word forms in the RSR condition than those in the repeated study condition; past studies have not consistently shown an advantage for recall of "meaning" or for recognition. It is also expected that children with TD will remember more words overall than children with DLD. To the degree that the story format is more engaging for children, overall recall will be enhanced for both groups. Assuming that the results are replicated, it is hoped that the children's book reading format will prove amenable for use by teachers and speech-language pathologists who work with children with DLD.

ELIGIBILITY:
Inclusion Criteria:

* a significant deficit in language ability (language test score below cutoff for best sensitivity/specificity) or documented age-appropriate language ability.
* normal hearing
* no evidence of neurological damage or disease
* scores on tests of nonverbal intelligence above the intellectual disability range
* not within Autistic range on Autism screening test
* native English speaker (can be bilingual)

Exclusion Criteria:

* failed hearing screening
* known neurological damage or disease
* scores on tests of nonverbal intelligence below the intellectual disability range (standard score less than 75)
* autism spectrum disorder
* non-native English speaker

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence B. Leonard, PhD, Principal Investigator — Purdue Universtiy
Locations (2):
- United States (2):
  - Purdue University's SLHS laboratories (8445 Keystone Crossing), Indianapolis, Indiana
  - Purdue University, West Lafayette, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Data that contribute to our final published results will be made available at clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after the results are published or within 12 months from the primary completion date (i.e., the date of final data collection for the primary outcome measure).
Access Criteria: De-identified data will be made publicly available at clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with DLD are recruited primarily through speech pathologists and preschool teachers. They are provided with eligibility guidelines and a parent letter. Once the parent is given the letter, they choose to contact us, if interested.
  Children with typical language development are recruited through advertising in preschools.
Pre-assignment Details: Children are initially tested to see if they meet the inclusionary and exclusionary criteria of Developmental Language Disorder. These include falling below age level on a language test, while passing a hearing screening, a non-verbal IQ test, and an autism screener. Many children who are recruited and consented do not meet all these criteria pointing to the fact that DLD is not readily recognizable to non-professionals (parents, preschool teachers).
Period: Overall Study
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.13 (7.57) | 57.07 (6.76) | 58.06 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 12 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Maternal Education in Years [Mean (Standard Deviation); unit: years] | 17.23 (3.77) | 18.04 (2.31) | 17.39 (3.24)

OUTCOME MEASURES:

1. Primary Outcome: Word Form Accuracy (Number of Words Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 5 Mins.
Description: Five minutes after second learning session, the child was asked to recall and say the word associated with each novel referent, learned under one of two conditions: a condition in which spaced retrieval trials occurred (RSR) and one in which there were no retrieval trials (RS). Each of the four verbs were tested twice, for a total of 8 recall items per condition.
Time Frame: 5 minutes after end of learning period
Measure: Mean (Standard Error); unit: number of words correctly recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 13 | 14
number of words correctly recalled
  RSR condition | 4.54 (0.58) | 6.5 (0.56)
  RS condition | 1.46 (0.59) | 4.0 (0.56)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p < 0.00001, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.00001, LSD test

2. Primary Outcome: Word Form Accuracy (Number of Words Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 1 Week.
Description: One week after second learning session, the child was asked to recall and say the word associated with each novel referent, learned under one of two conditions: a condition in which spaced retrieval trials occurred (RSR) and one in which there were no retrieval trials (RS). Each of the four verbs were tested twice, for a total of 8 recall items per condition.
Time Frame: 1 week after end of learning period
Measure: Mean (Standard Error); unit: number of words correctly recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 13 | 14
number of words correctly recalled
  RSR | 3.92 (0.70) | 6.07 (0.67)
  RS | 1.46 (0.52) | 3.43 (0.50)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p < 0.00001, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.00001, LSD test

3. Primary Outcome: Word Meaning Recall Accuracy (Number of Semantic Associations Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 5 Mins.
Description: Five minutes after second learning session, the child was asked to recall and say the semantic information associated with each novel referent, learned under one of two conditions: a condition in which spaced retrieval trials occurred (RSR) and one in which there were no retrieval trials (RS). Each of the four verbs were tested twice, for a total of 8 recall items per condition.
Time Frame: 5 minutes after end of learning period
Measure: Mean (Standard Error); unit: number of meanings correctly recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 13 | 14
number of meanings correctly recalled
  RSR | 7.31 (0.42) | 7.50 (0.40)
  RS | 5.46 (0.55) | 5.71 (0.53)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p < 0.00001, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.00001, LSD test

4. Primary Outcome: Word Meaning Recall Accuracy (Number of Semantic Associations Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 1 Week.
Description: One week after second learning session, the child was asked to recall and say the semantic information associated with each novel referent, learned under one of two conditions: a condition in which spaced retrieval trials occurred (RSR) and one in which there were no retrieval trials (RS). Each of the four verbs were tested twice, for a total of 8 recall items per condition.
Time Frame: 1 week after end of learning period
Measure: Mean (Standard Error); unit: number of meanings correctly recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 13 | 14
number of meanings correctly recalled
  RSR | 6.77 (0.40) | 7.21 (0.39)
  RS | 5.23 (0.52) | 5.57 (0.50)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p < 0.0001, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.00001, LSD test

5. Primary Outcome: Word Recognition (Number of Words Accurately Identified) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions.
Description: Upon hearing a novel word, the child is asked to indicate (by pointing) which picture among 3 options is referred to; for words learned under the RSR and RS conditions.
Time Frame: 1 week after end of learning period
Measure: Mean (Standard Error); unit: number or words correctly recognized
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 13 | 14
number or words correctly recognized
  RSR | 6.92 (0.32) | 7.86 (0.31)
  RS | 6.46 (0.25) | 7.86 (0.24)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p = 0.17, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p = 1.00, LSD test

6. Secondary Outcome: Peabody Picture Vocabulary Test, Fourth Edition
Description: The Peabody Picture Vocabulary is an individually administered, norm-reference test that assesses receptive vocabulary (ability to understand individual words) for children and adults ages 2 years 6 months to 90 years and older. Standard scores are derived from number correct. Standard scores can range from a minimum of 40 and 160. Standard scores between 85 and 115 (1 standard deviation above and below the mean of 100) are interpreted as reflecting receptive vocabulary levels expected for age. Scores below 85 are interpreted as reflecting receptive vocabulary levels below what is expected for age.Scores above 115 are interpreted as reflecting receptive vocabulary levels above what is expected for age.
Time Frame: Test completed at start of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 13 | 14
score on a scale | 100 (10.20) | 121.57 (10.60)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder vs Children With Typical Language Development; Test type: Superiority; p < 0.0001, LSD test

7. Secondary Outcome: Years of Maternal Education
Description: Educational attainment of child's mother in terms of years of education
Time Frame: Information collected at start of study
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 13 | 14
Years | 17.23 (3.77) | 18.04 (2.31)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder vs Children With Typical Language Development; Test type: Superiority; p = 0.51, LSD test

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT06026124/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT06026124/ICF_002.pdf